CLINICAL TRIAL: NCT01763502
Title: The Impact of Cash and Food Transfers Linked to Preschool Enrollment on Child Nutrition and Cognitive Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: United Nations World Food Programme (WFP) (Other); UNICEF (Other)
Responsible Party: Principal Investigator, Shalini Roy, Postdoctoral fellow, Poverty Health and Nutrition Division, International Food Policy Research Institute
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1004649
Record Dates: First submitted 2013-01-03; First posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Cognitive Development; Anemia
Keywords: Cognitive development; Anemia; Preschool; Food transfers; Cash transfers; Early childhood; Nutrition
MeSH Terms: conditions — Anemia | interventions — Food

ARMS (3):
- FOOD (Experimental): Food transfer linked to preschool enrollment
  Interventions: Other: FOOD
- CASH (Experimental): Cash transfer linked to preschool enrollment
  Interventions: Other: CASH
- CTRL (No Intervention): No transfer linked to preschool enrollment

INTERVENTIONS:
Other: FOOD — The food transfers consist of multiple-micronutrient-fortified corn soy blend (CSB), oil, and sugar, totaling approximately 1200 calories per day per child and including 99% of iron requirements.
  Arms: FOOD
Other: CASH — Cash transfers equal the estimated value of the food basket if purchased in the market.
  Arms: CASH

SUMMARY:
Recent evidence shows that early childhood is a critical period for investments in human capital and that micronutrient deficiency and inadequate stimulation are major causes of impaired child development in poor countries. These findings have increased interest in promoting nutrition interventions and preschool participation during early childhood. Transfers to households linked to preschool participation have the potential to improve nutrition and cognitive outcomes in young children. Receipt of transfers may induce improvements in diet quality and greater preschool participation, enhancing both nutrition and stimulation. However, there is limited evidence on the impacts of such programs, all of it from Latin America. There is also no evidence on the relative impact of different transfer modalities linked to preschool participation.

This study is a cluster-randomized controlled evaluation of a transfer program linked to preschool participation. The transfer program, administered by the World Food Programme, provides food or cash transfers to children aged 3-5 years enrolled in preschools at baseline. The preschools, operating in the Karamoja sub-region of Uganda, are supported by UNICEF and managed by District representatives of the Government of Uganda. The food transfers consist of multiple-micronutrient-fortified corn soy blend (CSB), oil, and sugar, totaling approximately 1200 calories per day per child and including 99% of iron requirements. Cash transfers equal the estimated value of the food basket if purchased in the market. Randomization into the food treatment, cash treatment or control was done across 98 preschools, referred to as Early Childhood Development (ECD) centers. The intervention period was from February 2011 to May 2012 and included distribution of transfers on a six-to-eight-week cycle. A longitudinal (panel) survey of households with children aged 3-5 years at baseline was conducted before exposure to the transfers and 18 months later. The randomized design of this effectiveness study and the panel nature of the data allow for a rigorous field trial in which impacts on nutrition and cognitive outcomes can be assessed and compared across modalities.

We examine the impacts of the two transfer modalities, cash transfers or multiple-micronutrient-fortified food transfers, linked to preschool enrollment, on child nutrition and cognitive development. In addition, we explore potential mechanisms through intermediate impacts on food intake and participation in preschools.

The key research objectives are to assess the following:

1. Impacts on targeted groups: Assess the effects of cash or food transfers on nutrition and cognitive outcomes in children aged 3-5 years at baseline and explore pathways for these effects.
2. Optimal program design: Assess the differential impacts of a program in which children are provided multiple-micronutrient-fortified food transfers linked to preschool enrollment compared with one in which they are given the equivalent value of cash transfers linked to preschool enrollment.

DETAILED DESCRIPTION:
Allocation: Randomized

This evaluation is conducted in communities surrounding Early Childhood Development (ECD) centers in the Karamoja sub-region of Uganda, in Napak, Kotido, and Kaabong districts. The catchment area of ECD centers serve as the clusters for randomization and analysis. After stratifying ECD centers (by district for Napak and Kotido, and by sub-district for the more spatially-diverse Kaabong), clusters were assigned to the treatment groups (FOOD, CASH and CTRL) using block randomization, to ensure as equal a distribution of ECD centers across treatment arms within each stratum as possible. Block randomization yielded 33 ECD centers in the FOOD group, 32 centers in the CASH group, and 33 centers in the CTRL group. Subsequently but prior to the start of the interventions, WFP re-assigned one CTRL center to FOOD, due to its proximity to a nearby FOOD center, in order to avoid migration of children which posed contamination concerns. WFP also re-assigned one CASH center to FOOD, because the cash distribution systems required use of mobile phones, and mobile phone signals were not readily available in the center's catchment area. The final assignment included 35 ECD centers in the FOOD group, 31 centers in the CASH group, and 32 centers in the CTRL group.

Statistical Analysis:

* Sample Selection and Sample Size: Prior to the baseline survey, power calculations were conducted using existing data from Uganda on cognitive measures (Mullens scores) and food security measures (share of food expenditures out of total expenditures) to estimate the necessary sample size for detecting a minimum effect size of 10 percentage points with 80 percent power. These calculations indicated a target minimum sample of 30 ECD centers per treatment arm and 20 households per ECD center. 98 ECD center clusters were determined eligible for transfer receipt by WFP. ECD enrollment data collected in August-September, 2010, were used to identify households with children ages 3-5 years enrolled in these ECD centers. In each of the 98 ECD centers, out of all households with children ages 3-5 years enrolled, roughly 25 households were selected at random for inclusion in the baseline sample.
* Data Collection: The evaluation uses a longitudinal design, with the same households interviewed at baseline (September-November, 2010, prior to start of the food or cash program) and at endline (March-May, 2012). In the intervening months, treatment households receive 15 months of exposure to the intervention. Direct assessments of children's cognitive development, anthropometry, and hemoglobin levels are conducted in a randomly-selected roughly 80% of sampled households in each cluster, due to field time constraints. Cognitive development is assessed using a battery of test items drawn primarily from the Mullen Scales of Early Learning, adapted by psychologists for the Karamoja context. Anthropometry is measured following standard protocol using height boards and weighing scales. Hemoglobin concentration is assessed using capillary blood obtained by finger prick and read using a HemoCue® analyzer. Hemoglobin readings are adjusted as necessary for the effects of varying altitude in the sample.
* Analysis: Differences in baseline characteristics are assessed using pairwise t-tests and binomial probability tests. Analyses of impacts focus on outcomes for children age 3-5 years (36-71 months) at baseline, as well as for children aged 36-53 months at baseline who remain in the targeted age range throughout the course of the intervention. Intent to treat (ITT) effects are estimated using single-difference and ANCOVA specifications on children at baseline and endline. Estimates are calculated using Stata 12; standard errors account for stratification and clustering in sampling and assignment.

Ethics Review:

* Side Effects: Potential risks from participation in this study are low. Many of the questions used in the survey have been used before in the Uganda National Household Survey. Cognitive tests consist of simple games played between a trained enumerator and the child and are unlikely to pose any risk to the children. Anthropometry measurements are non-invasive and also pose no risk. Risks associated with hemoglobin data collection are minimized through use of well-trained staff, a well-designed data collection protocol, and safety lancets. The study poses no social, emotional, or psychological risks to subjects.
* Health provisions: If any child is found to be severely anemic (Hb<7 g/dL) or wasted (weight-for-height less than two standard deviations below the mean), that child and the child's parents are notified and the child is referred to the nearest clinic for medical treatment.
* Informed consent: Details about the study are provided verbally to local leaders at the LC1 (roughly the equivalent of a village) level. The same information, including the right to opt out at any time, is provided verbally to survey respondents in sampled households. Additional informed consent is sought before each direct interaction with children, including for cognitive tests, anthropometry, and hemoglobin measurement.
* IRB: This study underwent internal review with the International Food Policy Research Institute; permission to conduct the data collection was granted by Uganda National Council for Science and Technology (SS 2470).

Funding:

This evaluation was funded by the World Food Programme, with support from the Spanish government and other sources through the Strategic Impact Evaluation Trust Fund at WFP, and by the United Nations Children's Fund.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3-5 years
* Enrolled in ECD centers funded by UNICEF at baseline

Exclusion Criteria:

* None

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2561 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Cognitive development scores at 18 months after baseline | March-May, 2012: 18 months after baseline
  Mullens total raw score, visual reception domain score, fine motor domain score, receptive language domain score, expressive language domain score
Anemia incidence at 18 months after baseline | March-May, 2012: 18 months after baseline
  Mild anemia (hemoglobin concentration < 11•0 g/dL); moderate to severe anemia (hemoglobin concentration < 9•0 g/dL)

SECONDARY OUTCOMES:
Anthropometry at 18 months after baseline | March-May, 2012: 18 months after baseline
  Prevalence of stunting; prevalence of underweight; prevalence of wasting

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Gilligan, PhD, Principal Investigator — International Food Policy Research Institute; Shalini Roy, PhD, Principal Investigator — International Food Policy Research Institute
Locations (1):
- UNICEF early childhood development centers, Karamoja Sub-region, Uganda